CLINICAL TRIAL: NCT02425462
Title: EffectiveNess of VISanne® in Improving Quality of Life in asIan wOmen With eNdometriosis
Brief Title: To Evaluate Effectiveness of Visanne in Improving Quality of Life in Asian Women With Endometriosis
Acronym: ENVISIOeN
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17444
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — dienogest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Asian patients at least 18 years of age with clinical or surgical diagnosis of endometriosis, and patients with endometriosis associated pelvic pain.
  Interventions: Drug: Dienogest (Visanne, BAY86-5258)

INTERVENTIONS:
Drug: Dienogest (Visanne, BAY86-5258) — Dienogest 2mg daily Oral dose

SUMMARY:
This study is a prospective observational cohort study. The study will be conducted in routine clinical practice settings. It is planned to enroll 870 patients with endometriosis for whom a decision has been made by the physician to treat with dienogest according to local health authority approved label. It is the aim of this observational cohort study to further characterize the effectiveness of dienogest in improving quality of life and long-term safety in routine clinical practice setting. Endometriosis is chronic and progressive disease and there is unmet need for long-term treatment. Visanne® with proven efficacy and safety, can be good option for long-term treatment, however, experience with Visanne® beyond 15 month is limited. And long-term up to 24 months data on effectiveness and safety of Visanne would support the long-term treatment strategy for Endometriosis management in the clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Asian Female patients at least 18 years of age
* Clinical or surgical diagnosis of endometriosis (depending on local approved indication) : Clinical diagnosis by suggestive symptoms and positive finding in imaging study (Chocolate cyst)
* Patients with Endometriosis associated pelvic pain
* Decision taken by the physician to newly prescribe Visanne®
* Availability of a signed informed consent

Exclusion Criteria:

* Patients participating in an investigational program with interventions outside of routine clinical practice
* Patients for whom any of contraindication listed in the local summary of product characteristics (SPC) apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asian patients at least 18 years of age with Clinical or surgical diagnosis of endometriosis, and patients with endometriosis associated pelvic pain
Sampling Method: Probability Sample
Enrollment: 895 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
The mean change from baseline to 6 months of treatment in pain-related Quality of Life measured by EHP-30. | Baseline and at 6 months
The mean change from baseline to 24 months of treatment in pain-related Quality of Life measured by EHP-30 for patients who continue to take Visanne up to 24 months. | Baseline and to 24 months

SECONDARY OUTCOMES:
Mean change from baseline to 6 months and baseline to 24 months of treatment in other domain of Quality of life measured by EHP-30 | Baseline and 6 months,Baseline to 24 months
  Other domain includes control and powerlessness, emotional wellbeing, social support, self-image as well as modular domain including work life, sexual intercourse, relationship with children, treatment and concern on infertility
Mean change of Endometriosis-associated pelvic pain (EAPP) from baseline in patients with endometriosis either surgically or clinically diagnosed. | Baseline and 6 months, Baseline and 12 months, Baseline and 24 months
Patient and physician's satisfaction score on Visanne® treatment | At 6 months, 12 months, 24 months
  The subject and physician will be asked to choose any of following; very satisfied, somewhat satisfied, neither satisfied or dissatisfied, somewhat dissatisfied, very dissatisfied.
Proportion of subjects who continue treatment with Visanne® | At 6 months, 12 months, 24 months
Reasons for stopping of treatment with Visanne® | At 6 months, 12 months, 24 months
Proportion of patients with amenorrhea, intermenstrual bleeding/spotting or irregular bleeding while treatment with Visanne® | At 1 month, 3 months, 6 months, 12 months, and 24 months
Proportion of patients who experienced pain recurrence in patients taking Visanne up to 24 months | Up to 24 months
Time point for first pain recurrence after stopping taking Visanne and before to start any treatment. | Up to 24 months
  Pain recurrence is defined as severity of pain graded > 4 on the 10-point NRS
Proportion of patients who underwent repeated surgery in patients taking Visanne up to 24 months | Up to 24 months
Proportion of patients who underwent repeated surgery between stopping Visanne treatment and starting any other treatment than surgery | Up to 24 months
Patient's assessment of overall symptom development using the Clinical Global Impression (CGI) scale | At 6 months, 12 months, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- Multiple Locations, Indonesia
- Multiple Locations, Malaysia
- Multiple Locations, Philippines
- Multiple Locations, Singapore
- Multiple Locations, South Korea
- Multiple Locations, Thailand

REFERENCES:
- [Result] Techatraisak K, Hestiantoro A, Ruey S, Banal-Silao MJ, Kim MR, Seong SJ, Thaufik S, Ahlers C, Shin SY, Lee BS. Effectiveness of dienogest in improving quality of life in Asian women with endometriosis (ENVISIOeN): interim results from a prospective cohort study under real-life clinical practice. BMC Womens Health. 2019 May 16;19(1):68. doi: 10.1186/s12905-019-0758-6. PMID 31096979
- [Derived] Techatraisak K, Hestiantoro A, Soon R, Banal-Silao MJ, Kim MR, Seong SJ, Hidayat ST, Cai L, Shin S, Lee BS. Impact of Long-Term Dienogest Therapy on Quality of Life in Asian Women with Endometriosis: the Prospective Non-Interventional Study ENVISIOeN. Reprod Sci. 2022 Apr;29(4):1157-1169. doi: 10.1007/s43032-021-00787-w. Epub 2022 Feb 2. PMID 35112299